CLINICAL TRIAL: NCT07401290
Title: The Safety and Efficacy of Direct SLT in Pseudoexfoliation Glaucoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vance Thompson Vision (Other)
Responsible Party: Principal Investigator, Lorraine Provencher, Sponsor-Investigator, Vance Thompson Vision
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSLT_PXFG IIT
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pseudoexfoliation Glaucoma
MeSH Terms: conditions — Exfoliation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treated Group (Experimental): Patients treated with DSLT
  Interventions: Device: Direct selective laser trabeculoplasty

INTERVENTIONS:
Device: Direct selective laser trabeculoplasty — A non-invasive laser procedure for treating glaucoma and ocular hypertension by improving the eye's natural fluid drainage

SUMMARY:
Prospective, multi-center, single arm, interventional study evaluating DSLT in patients with pseudoexfoliative glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with pseudoexfoliation glaucoma (PXFG), with optic neuropathy consistent with glaucomatous damage of any severity
* Open iridocorneal angle by gonioscopy, defined as a Shafer Grade II or greater
* Treatment naive, or washed out IOP ranging from ≥18-35 mmHg
* Able to complete medication washout safely and all follow-up visits
* Participants must have a best correct visual acuity of 20/40 or better in the study eye(s), be able to undertake a reliable Humphrey visual field (HVF) (defined as fixation losses, false positives and false negatives less than 33%), and must have field loss no worse than -20 dB in treatment eye

Exclusion Criteria:

* Any contraindication to SLT or unable to have DSLT
* Angle closure glaucoma or any other types of glaucoma other than PXFG
* Prior incisional glaucoma surgery or glaucoma-related procedures in the study eye
* Any prior refractive surgery
* H/o LPI within last 6 months
* A history of any significant cataract required during study duration or cataract surgery in the last 6 months
* Prior laser trabeculoplasty (ALT/SLT)
* History of ocular inflammation and infection
* Patients who are pregnant or have any clinically relevant systemic disease that may prevent them from reliably completing follow-up visits
* Vulnerable populations that cannot provide proper informed consent will not be enrolled, such as children, prisoners, handicapped, or mentally disabled persons, or economically or educationally disadvantaged persons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Primary Effective Endpoint | 6 months
  Proportion of eyes achieving ≥20% reduction in washed-out IOP at month 6 compared to washed-out baseline IOP

SECONDARY OUTCOMES:
Secondary Effective Endpoint | 12 months
  Proportion of eyes achieving ≥ 20% reduction in washed out IOP at month 12 compared to washed-out baseline IOP
Secondary Effective Endpoint | 6 and 12 months
  Mean washed out IOP reduction at 6 and 12 months as compared to washed-out baseline IOP
Secondary Effective Endpoint | 6 and 12 months
  Change in # of glaucoma medication(s) at 6 and 12 months
Secondary Effective Endpoint | 6 and 12 months
  Proportion of medication free eyes post-DSLT at 6 and 12 months
Secondary Effective Endpoint | 12 months
  Rate of secondary surgical interventions (SSIs) at 12 months
Secondary Effective Endpoint | 12 months
  Kaplan-Meier survival analysis at 12 months: time to failure (failure defined as an increase in glaucoma medications from baseline or additional IOP lowering procedure)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Vance Thompson Vision, Alexandria, Minnesota
  - Vance Thompson Vision, Omaha, Nebraska
  - Vance Thompson Vision, Fargo, North Dakota